CLINICAL TRIAL: NCT02714842
Title: A Pharmacoscintigraphic Clinical Study to Investigate the in Vivo Behaviour of a Novel Delayed-release Formulation of Diclofenac in Comparison to the Voltaren® Enteric Coated Tablet Commercial Formulation in Healthy Volunteers
Brief Title: Delayed Release Diclofenac Sodium Formulation vs Voltaren®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BDD Pharma Ltd (Industry)
Collaborators: Drug Delivery International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: FM1501
Record Dates: First submitted 2016-03-08; First posted 2016-03-22 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Radiolabelled Diclofenac tablet A (Experimental): Single dose of delayed release diclofenac sodium (50 mg) tablet radiolabelled with 4 MBq 99mTc
  Interventions: Drug: Radiolabelled Diclofenac Tablet A
- Radiolabelled diclofenac tablet B (Experimental): Single dose of delayed release diclofenac sodium (50 mg) tablet radiolabelled with 4 MBq 99mTc
  Interventions: Drug: Radiolabelled Diclofenac tablet B
- Voltaren (Active Comparator): Single dose of enteric coated diclofenac sodium (50 mg) tablet radiolabelled with 4 MBq 99mTc
  Interventions: Drug: Diclofenac
- Radiolabelled diclofenac tablet C (Experimental): Single dose of delayed release diclofenac sodium (25 mg) tablet radiolabelled with 4 MBq 99mTc
  Interventions: Drug: Radiolabelled Diclofenac tablet C

INTERVENTIONS:
Drug: Radiolabelled Diclofenac Tablet A — Delayed release diclofenac sodium tablet (50 mg)
  Other Names: Delayed release diclofenac sodium tablet
  Arms: Radiolabelled Diclofenac tablet A
Drug: Radiolabelled Diclofenac tablet B — Delayed release diclofenac sodium tablet (50 mg)
  Other Names: Delayed release diclofenac sodium tablet
  Arms: Radiolabelled diclofenac tablet B
Drug: Radiolabelled Diclofenac tablet C — Delayed release diclofenac sodium tablet (25 mg)
  Other Names: Delayed release diclofenac sodium tablet
  Arms: Radiolabelled diclofenac tablet C
Drug: Diclofenac — Enteric coated delayed release diclofenac sodium tablet (50 mg)
  Other Names: Voltaren
  Arms: Voltaren

SUMMARY:
This is a single-centre, open-label, randomised, three-arm crossover study with a fourth fixed arm in a subset of subjects. Up to 36 healthy male volunteers will participate in the study. This study is designed to correlate the gastrointestinal transit behaviour of delayed-release diclofenac sodium tablets with their pharmacokinetic (PK) absorption profiles.

The investigators will be looking at:

1. The behaviour of the tablets (when, where and how quickly they break up)
2. The gastric emptying time of the tablets (when they leave the stomach)
3. The gastrointestinal transit of the tablets (how long they take to travel through the gut)
4. Blood levels of the drug (diclofenac)

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 18 and 55 years inclusive.
* Weight & Body mass index (BMI)
* BMI between 18.0 and 29.9 kg/m², inclusive. Body weight ≥50 kg
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* Good general health with (in the opinion of the Investigator) no clinically significant and relevant abnormalities of medical history or physical examination.

Exclusion Criteria:

* Current or relevant previous history of severe or uncontrolled disease that, in the opinion of the physician responsible, could affect the study conduct or laboratory assessments (e.g., renal, cardiovascular, hepatic, hematologic, endocrine, pulmonary, psychiatric, neurologic, or cerebral disease).
* Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.
* A history of current or relevant previous non self-limiting gastrointestinal disorders in particular, peptic ulcer disease and/or gastrointestinal bleeding.
* A history of hypersensitivity to aspirin or any other NSAID.
* Suffering from asthma requiring current treatment.
* Currently suffering from disease known to impact gastric emptying, e.g., migraine, insulin-dependent diabetes mellitus.
* Laboratory screening results that suggest an abnormal liver and/or renal function.
* Subject has a screening QTc value of greater than or equal to 450 msec or an ECG that is not suitable for QTc measurements (e.g., poorly defined termination of the T-wave). The ECG taken at screening must be considered not clinically significant by the Investigator/ study physician.
* Currently suffering from bleeding or coagulation disorders.
* As a result of a physical examination or screening investigations, the physician responsible considers the volunteer unfit for the study.
* Subject has taken prescribed medication within 14 days prior to the first assessment visit which, in the opinion of the physician responsible, will interfere with the study procedures or compromise safety. Subjects will be withdrawn from subsequent study days if they commence taking prescribed medication during the study period which, in the opinion of the physician responsible, will interfere with the study procedures or compromise safety.
* Subject has taken over-the-counter (OTC) medication within 48 hours prior to each assessment visit. T This includes the use of vitamins and natural or herbal remedies e.g., St John's Wort. Subjects who have taken OTC medication may still be entered into the study if, in the opinion of the physician responsible, the medication will not interfere with the study procedures or compromise safety. The occasional use of paracetamol for pain relief (within its labelled dosage) is permitted but must not be taken within 48 hours of an Assessment Visit.
* Recent history (within the last year) of alcohol or other substance abuse.
* Subject has an average weekly alcohol intake of greater than 21 units. 1 unit is equivalent to one 25 mL single measure of whisky, or a third of a pint of beer or half a standard (175 mL) glass of red wine.
* Subject has positive urine drugs of abuse test at screening. Note: At the discretion of the Investigator, the test may be repeated.
* Subject has a positive breath alcohol test at screening.
* Subject has recently discontinued smoking (less than 3 months).
* Subject is currently a smoker or user of nicotine-containing products.
* Subject has a history of allergy to the study drug diclofenac sodium, to any component of the dosage form or any other allergy, which, in the opinion of the physician responsible, contraindicates their participation.
* Has an allergy to any of the contents of the meals.
* Subject is vegetarian.
* Subject claims to be lactose intolerant.
* Participation in another clinical study (inclusive of final post-study examination) or receipt of an investigational drug within the 12 weeks before screening visit.
* Previous participation in this study.
* Subject whose participation in this study will result in a participation in more than four studies over a twelve month period.
* An employee of the sponsor, client or study site or members of their immediate family.
* Subjects for whom participation in this study will exceed the limits of total radiation exposure allowed in any 12 month period (5 mSv), or will exceed 10 mSv over any three year period.
* Subjects who are intending to father a child in the 3 months following the study or are unwilling to abstain from sexual intercourse with pregnant or lactating women.
* Subjects who are unwilling to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first assessment visit until 3 months following the study.
* Subject has donated blood or experienced significant blood loss within 3 months of screening and throughout the duration of the study.
* Difficulty accessing forearm veins for cannulation or blood sampling.
* Subject has any non-removable metal objects such as metal plates, screws etc. in their chest or abdominal area.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal transit parameters - gastric emptying time, small intestinal transit time, and colon arrival time of radiolabel where applicable. | 16 hours
  Composite outcome

SECONDARY OUTCOMES:
Scintigraphic analysis to determine the times and sites of onset and complete release of radiolabelled lactose. | 16 hours
  Composite outcome
Pharmacokinetic parameters plasma concentration (Cp) at each PK sampling point. | 20 hours

CONTACTS AND LOCATIONS:
Overall Officials: Howard NE Stevens, Principal Investigator — BDD Pharma Ltd
Locations (1):
- Bio Images Research Ltd, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No